CLINICAL TRIAL: NCT02396355
Title: Accuracy Evaluation of the BD FACS Presto System: Instrument, Software and BD CD4/%CD4/Hb Cartridge Assay
Brief Title: Accuracy Evaluation of the BD FACS Presto System
Status: Completed | Type: Observational
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CAS-PCACC1
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Acquired Immunodeficiency Syndrome
Keywords: flow cytometry
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All subjects: This is a single arm study. Samples from each subject will be tested with the Investigational BD FACSPresto System, the BD FACSCalibur flow cytometer, and the Sysmex hematology analyzer KX-21.
  Interventions: Device: Investigational BD FACSPresto System; Device: BD FACSCalibur flow cytometer; Device: Sysmex hematology analyzer KX-21

INTERVENTIONS:
Device: Investigational BD FACSPresto System — Blood samples will be tested on the BD FACSPresto system for CD4 absolute count (CD4Abs), %CD4, and Hb concentration.
Device: BD FACSCalibur flow cytometer — Blood samples will be tested on the predicate, currently marketed device. For CD4Abs and %CD4 measurement, the BD FACSCalibur flow cytometer will be used with BD Multiset software version 1.1 or later and BD Tritest CD3/CD4/CD45 reagent with Trucount tubes.
Device: Sysmex hematology analyzer KX-21 — Blood samples will be tested for hemoglobic concentration on the predicate, currently marketed Sysmex hematology analyzer KX-21

SUMMARY:
The enumeration of T lymphocytes positive for the CD4 antigen is used to determine the immune status of patients with, or suspected of developing, immune deficiencies such as AIDS. The BD FACS Presto™ is an investigational automated system for in vitro diagnostic use in performing the direct enumeration of CD4 absolute count, CD4 percentage of lymphocytes, and hemoglobin (Hb) concentration in human whole blood.

This is a prospective study to determine the relative bias between the investigational BD FACS Presto system and the predicate BD FACS Calibur with BD Tritest system in their determination of absolute CD4, % CD4, and Hb concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been infected with HIV and willing to provide informed consent to draw venous and capillary blood
* Specimen: Venous blood must be collected in blood collection tube with EDTA anticoagulant and stored at room temperature (20-25 °C) according to tube manufacturer's instructions
* Specimen: post enrolment staining within 24 hours
* venous blood of acceptable quality for flow cytometry, e.g. no hemolysis or clots and acceptable pre analytical handling)
* venous blood sample > 1 mL for sample preparation
* capillary blood applied to the investigational CD4/%CD4/Hb cartridge

Exclusion Criteria:

* Subject unwilling to disclose medical information regarding previous CD4 test results
* Subject unwilling to discuss medical information regarding co-morbid conditions and current medications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll specimens from children 0-12 years and adolescent or adult patients 13 years of age or greater. Enrolment of children in the study is expected to satisfy the binning (stratification) requirements since relative lymphocytosis and higher CD4+ lymphocyte counts are normal in children less than 5 years of age.
Enrollment: 583 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Method bias between BD FACSPresto System vs. Predicate in venous blood (AbsCD4 and %CD4) | assayed upon sample collection
  The primary endpoint is the bias (expected difference) between the investigational vs. predicate system measured as absolute CD4 lymphocyte count and %CD4 in peripheral venous blood from a minimum of 400 specimens with valid results tested at three or more external sites.

SECONDARY OUTCOMES:
Method bias between BD FACSPresto System vs. Predicate in Capillary Blood (AbsCD4 and %CD4) | assayed upon sample collection
  The bias (expected difference) between the investigational vs. predicate system measured as absolute CD4 lymphocyte count and %CD4 in capillary blood from a minimum of 400 specimens with valid results tested will be determined at three or more external sites.
Method bias between BD FACSPresto System vs. Predicate for Hemoglobin | assayed upon sample collection
  The bias (expected difference) between the investigational BD FACSPresto system vs. predicate (Sysmex KX-21 hematology analyzer) will be determined for hemoglobin concentration using venous blood and capillary blood.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Judge, MD, Study Chair — Becton, Dickinson
Locations (6):
- United States (3):
  - Children's Hospital Los Angeles, Los Angeles, California
  - San Francisco General Hospital and Trauma Center, San Francisco, California
  - Becton Dickinson MedLab, San Jose, California
- National AIDS Research Institute, Pune, Maharashtra, India
- KEMR/CDC Research and Public Health Collaboration, Kisumu, Kenya
- Siriraj Hospital, Bangkok, Siriraj, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Angira F, Akoth B, Omolo P, Opollo V, Bornheimer S, Judge K, Tilahun H, Lu B, Omana-Zapata I, Zeh C. Clinical Evaluation of the BD FACSPresto Near-Patient CD4 Counter in Kenya. PLoS One. 2016 Aug 2;11(8):e0157939. doi: 10.1371/journal.pone.0157939. eCollection 2016. PMID 27483008